CLINICAL TRIAL: NCT05826990
Title: Single Group Phase 2 Study to Investigate Pharmacokinetics, Safety and Tolerability of Cefepime-Enmetazobactam Administered by IV Over 2 Hr in Male or Female Participants From Birth to Less Than 18 Years of Age Hospitalised With cUTI
Brief Title: A Study to Investigate PK, Safety, Tolerability of Cefepime-enmetazobactam in Pediatric Participants With cUTI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Allecra (Industry)
Collaborators: Linical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-202
Record Dates: First submitted 2023-01-30; First posted 2023-04-24 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Complicated Urinary Tract Infection
MeSH Terms: interventions — Cefepime; cefepime, enmetazobactam drug combination

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- cefepime and enmetazobactam unique study arm (Experimental): Each study participant will receive a two-hour intravenous administration of cefepime and enmetazobactam every 8 hours, as single drug in fixed dose combination (FDC) formulation at a ratio of 4 to 1.
  Interventions: Drug: cefepime and enmetazobactam combination

INTERVENTIONS:
Drug: cefepime and enmetazobactam combination — Cefepime and enmetazobactam fixed dose combination administered intravenously every 8 hours as single drug formulation
  Other Names: cefepime-enmetazobactam

SUMMARY:
This phase 2 study is part of regulatory commitments in the United States (PSP) and Europe (PIP) to evaluate cefepime-enmetazobactam in paediatric participants with cUTI to support extension of the indication for cefepime-enmetazobactam to children with cUTI.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the blood concentrations and safety of the fixed dose combination of 2 drugs, cefepime with enmetazobactam administered intravenously in participants aged from birth to less than 18-years of age, hospitalised with a complicated urinary tract infection.

The treatment duration will be between 3 and 7 days, depending on the time needed for disappearance of signs and symptoms of the infection.

The participant will need to be hospitalised at least during the treatment administration period. After the last administration of cefepime and enmetazobactam, there will be the end of treatment visit (EOT), then 2 follow-up visits at 7 days (Test of Cure (TOC)), then 14 days (Late Follow-up (LFU)) after the end of treatment visit. The End of study Visit (EOS) will be conducted via telephone call (or a visit deemed necessary as per the investigator) 28 days after the EOT visit. The participants may be discharged from hospital at the discretion of the investigator after the end of treatment visit but will be required to return to the hospital for the 2 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be from birth to <18 years of age. Participants up to 2 months must have been born at term or preterm with a gestational age ≥32 weeks.
* Written informed consent from parent(s) or other legally acceptable representative(s), and informed assent from participant (if age appropriate according to local regulations).
* If female and has reached menarche, or has reached Tanner stage 3 development, (even if not having reached menarche) the participant is authorized to participate in this clinical study if the following criteria are met:

  1. Participant has a negative urine and/or serum human chorionic gonadotropin test at screening visit. As serum tests may miss an early pregnancy, relevant menstrual history, and sexual history, including methods of contraception, should be considered
  2. Participant agrees to avoid conception from the time of screening until 7 days after receipt of study intervention and agrees not to attempt pregnancy from the time of screening until 7 days after EOT with study intervention, and participant agrees to follow guidelines received regarding continuation of abstinence, initiation of abstinence or about allowed contraception, and
  3. Participant reports sexual abstinence for the prior 3 months or reported the use of at least 1 of the acceptable methods of contraception, including an intrauterine device (with copper banded coil), levonorgestrel intrauterine system or regular medroxyprogesterone injections, or participant agrees to initiate sexual abstinence from the time of screening until 7 days after end of treatment (EOT) with study intervention.
* Participant has a clinically suspected and/or bacteriologically documented complicated urinary tract infection (cUTI) or acute pyelonephritis judged by the investigator to require the participant to be hospitalized for treatment with intravenous (i.v.) therapy.
* The causative pathogen is confirmed or suspected to be susceptible to cefepime-enmetazobactam.
* Participant has pyuria, defined as dipstick analysis positive for leukocyte esterase OR:

  1. If ≥1 year of age: White blood cell (WBC) count >10 cells/µL in unspun urine or ≥10 cells/high power field in spun urine.
  2. If <1 year of age: WBC count >5 cells/µL in unspun urine or ≥5 cells/high power field in spun urine.
* Participant demonstrates clinical signs and/or symptoms of either acute pyelonephritis or cUTI at the Screening Visit, as defined by the following criteria:

  a. For pyelonephritis, participants must have at least 2 of the following new or worsening signs and/or symptoms: i. If 0 to <2 years of age:
  * Fever (as defined by the investigator)
  * Failure to thrive
  * Recent weight loss
  * Irritability
  * Poor feeding
  * Lack of normal level of activity
  * Abdominal tenderness on physical examination
  * Vomiting ii. If 2 to <18 years of age:
  * Fever (as defined by the investigator)
  * Dysuria
  * Urinary urgency
  * Urinary frequency
  * New-onset urinary incontinence
  * Suprapubic pain, flank pain, or abdominal pain
  * Suprapubic tenderness or CVA tenderness on physical examination
  * Nausea or vomiting OR

    b. For cUTI, participants must have at least 2 of the new or worsening signs and/or symptoms listed above AND must have at least 1 of the following complicating factors:
  * Obstructive uropathy
  * Congenital, functional, or anatomic abnormality of the urogenital tract
  * Temporary indwelling urinary catheter
  * Bladder instrumentation within <24 hours
  * Recurrent UTI (≥2 events within a 12-month period)
* Have a baseline urine culture specimen obtained within 48 hrs prior to the first dose of the study intervention. (Participants may be enrolled in this study and start i.v. study intervention therapy before the Investigator knows the results of the baseline urine culture in the event the causative pathogen is suspected to be susceptible to cefepime-enmetazobactam).

Specimen is to be obtained by suprapubic aspiration, clean intermittent urethral catheterization, indwelling urethral catheter, or mid- stream clean catch.

* Likely to survive the current illness or hospitalization.
* Sufficient intravascular access (peripheral or central) to receive study intervention

Exclusion Criteria:

* History of serious allergy, hypersensitivity (e.g., anaphylaxis), or any serious reaction to cefepime, any cephalosporin, penicillins, β-lactamase inhibitors (e.g., tazobactam, sulbactam, or clavulanic acid), or other β-lactam agents.
* Previous enrolment in this study, or in another interventional study ≤30 days before i.v. administration of study intervention.
* Concurrent infection requiring systemic antibiotics in addition to the i.v. study intervention therapy at the time of first study intervention administration.
* Receipt of systemic antibiotics within 24 hours before obtaining the study qualifying pre-treatment baseline urine sample and before study intervention therapy. Exceptions are:
* Receipt up to 24 hours of short-acting antibacterial agent with a daily dose not completed. (Refer protocol ► Section 10.5, Appendix 5 for the list of allowed and disallowed antibiotics).

  * Patients who received prior antimicrobial therapy for the current cUTI/AP, and 1) in the Investigator's opinion, failed that prior antibiotic therapy (i.e., presented with worsening signs and symptoms), AND 2) were documented that the pathogen is non-susceptible to the prior antibiotic therapy.
  * Patients who have received antimicrobial prophylaxis for recurrent cUTI and then presented signs and symptoms consistent with an active new cUTI or AP.
* A permanent indwelling bladder catheter or instrumentation including nephrostomy or current urinary catheter or anticipation of urinary catheter placement that would not be removed during the course of i.v. study intervention therapy administration.
* Participant has suspected or known complete obstruction of any portion of the urinary tract, perinephric abscess, or ileal loops.
* Participant has trauma to the pelvis or urinary tract.
* Participant has undergone renal transplantation.
* Participant has a condition or history of any illness that, in the opinion of the investigator, would have made the participant unsuitable for the study (e.g., may have confounded the results of the study or posed additional risk in administering the study therapy to the participant).
* Participant is considered unlikely to survive the 6-week study period or had a rapidly progressive illness, including septic shock, that was associated with a high risk of mortality.
* At the time of first study intervention administration, known presence of a cUTI caused by pathogens resistant to Cefepime - enmetazobactam.
* Presence of any of the following clinically significant laboratory abnormalities:

  1. Haematocrit <25% or haemoglobin <8 g/dL (<80 g/L, <4.9 mmol/L) for children ≥ 1 month, or <13 g/dL (<130 g/L, <8.0 mmol/L) for children < 1 month.
  2. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>3 times the age-specific upper limit of normal (ULN), or total bilirubin >2 times ULN (except known Gilbert's disease) and Absolute Neutrophil count<1000/ mm3.
  3. eGFR <30 mL/min/1.73m2. (updated creatinine-based "Bedside Schwartz" equation (Schwartz et al. 2009))
* Participant has baseline QTcB (corrected Bazett's formula) of greater than 450 msec.
* History of seizures, excluding well-documented febrile seizures of childhood.
* If female, currently pregnant or breast feeding.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics Cmax | Day 1 - Day 2
  Maximum Plasma Concentration [Cmax] ; unit= mg/L
Pharmacokinetics Tmax | Day 1 - Day 2
  Time to reach Cmax (Tmax) ; unit= h
Pharmacokinetics AUC0-tau | Day 1 - Day 2
  Area under the plasma concentration time curve from time zero to the end of the dosing interval (AUC0-tau) ; unit= mg.h/L
Pharmacokinetics AUC0-inf | Day 1 - Day 2
  Area under the concentration time curve from time zero extrapolated to infinity (AUC0-inf) ; unit= mg.h/L
Pharmacokinetics t1/2 | Day 1 - Day 2
  Elimination half-life (t1/2), apparent terminal elimination rate constant (λz) ; unit= h
Pharmacokinetics CL & Vd | Day 1 - Day 2
  Clearance (CL, volume of plasma cleared of the drug per unit time) ; unit= L, Volume of distribution (Vd) ; unit= L
Pharmacokinetics Cmin | Day 1 - Day 2
  Trough observed plasma concentration (Cmin) ; unit= mg/L
Safety and Tolerability | before 1st study intervention until EOT +28 Days (±5 Days)
  Patients with treatment emergent adverse events (AE); unit=percentage
Safety and Tolerability | before 1st study intervention until EOT +28 Days (±5 Days)
  Patients with drug related related treatment emergent (AE); unit=percentage
Safety and Tolerability | before 1st study intervention until EOT +28 Days (±5 Days)
  Patients with study intervention discontinuation due to AE; unit=percentage
Safety and Tolerability | before 1st study intervention until EOT +28 Days (±5 Days)
  Patients with serious adverse event (SAE); unit=percentage
Safety and Tolerability | before 1st study intervention until EOT +28 Days (±5 Days)
  Patients with drug related serious adverse event; unit=percentage

SECONDARY OUTCOMES:
Efficacy assessment | 7 Days (±2 Days) after the end-of-therapy (EOT)
  Efficacy Overall success rate (Combined clinical and microbiological success rate)
  * Clinical response
  * Microbiological response The main efficacy endpoint is the overall success rate (Combined clinical and microbiological success) in the m-MITT population at TOC.
  The other efficacy endpoints are listed below:
  * Clinical response of cure at TOC in m-MITT population
  * Microbiological response of eradication at TOC in m-MITT population
  * Overall success rate at Day 3, end-of-therapy (EOT), LFU in m-MITT population
  * Clinical response rate at the Day 3, EOT, LFU visits in m-MITT population
  * Microbiological response rate at the Day 3, EOT, LFU visits in m-MITT population
  * Overall success rate at Day 3, EOT, TOC, LFU in Clinically Evaluable (CE) and in microbiologically evaluable (ME) populations
  * Clinical response rate at Day 3, EOT, TOC, LFU in CE and ME populations
  * Microbiological response at the Day 3, EOT, LFU visits in CE and ME populations

CONTACTS AND LOCATIONS:
Locations (6):
- Fakultní nemocnice Hradec Králové -Ústav klinické biochemie a diagnostiky, Hradec Králové, Czechia
- Hopital des Enfants, Toulouse, France
- Debreceni Egyetem Klinikai Központ Gyermekgyógyászati Klinika, Debrecen, Hungary
- SZPZOZ im. Dzieci Warszawy w Dziekanowie Leśnym, Łomianki, Poland
- Národný ústav detských chorôb (NÚDCH), Bratislava, Slovakia
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No